CLINICAL TRIAL: NCT04801641
Title: Impact of Chronic Nabilone Self-administration on Body Weight, Metabolic Markers, Gut Microbiota, and Neural Circuitry in Human Obesity
Brief Title: A Pilot Trial of Nabilone for the Treatment of Obesity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor tolerability of medication and no preliminary efficacy
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 084/2018
Record Dates: First submitted 2021-03-04; First posted 2021-03-17 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Low-Dose Nabilone (Experimental): pms-nabilone titrated to 2 mg daily
  Interventions: Drug: Nabilone
- High-Dose Nabilone (Experimental): pms-nabilone titrated to 6 mg daily
  Interventions: Drug: Nabilone

INTERVENTIONS:
Drug: Placebo — Six placebo capsules taken orally twice daily
  Arms: Placebo
Drug: Nabilone — Titrated to two 0.5 mg capsules and four placebo capsules taken orally twice daily (Low-Dose) OR Titrated to six 0.5 mg capsules taken orally twice daily (High-Dose)
  Arms: High-Dose Nabilone; Low-Dose Nabilone

SUMMARY:
Obesity is a serious health problem which increases the likelihood of developing other life-changing medical conditions. Despite increasing knowledge about the neural and metabolic basis of obesity, the development of effective anti-obesity treatment strategies has been a challenge. Evidence shows an association between cannabis consumption and body weight. However, to date, no human trials have assessed the potential of cannabis-like compounds to reduce body weight in individuals who are obese. This pilot trial aims to determine the safety and feasibility of administering nabilone (a cannabinoid drug similar to the active component of cannabis) to patients who are obese. Our secondary aims are to determine if nabilone is effective in reducing weight in this population, and to probe potential mechanisms of the weight-loss-promoting effects of nabilone, such as neural reactivity to food stimuli, changes in gut bacteria, and changes in metabolic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Obese adults (BMI > 30.0 kg/m2).
* For the optional imaging component of the study, a maximum weight (315 lbs) and a maximum girth in line with capacity of the machine (60 cm horizontal and 45 cm vertical; therefore, circumference of scanner is 166.6 cm)
* For women of reproductive potential (WORP) and men whose sexual partners are WORP: use of adequate methods of contraception (effective barrier methods such as male condoms, female condoms, cervical caps, diaphragms, or contraceptive sponges; and highly effective methods of contraception such as oral hormonal contraceptives, intrauterine devices (IUDs), vasectomy, or tubal ligation)
* AST/ALT, bilirubin, and kidney function tests within normal limits at screening.

Exclusion Criteria:

* Unstable gastrointestinal, respiratory, endocrinological, cardiovascular or cerebrovascular diseases that would prevent participation in the trial at QI (or its delegate) discretion,
* Unstable major psychiatric disorder(s) (i.e. Axis I Disorders) that would prevent participation in the trial at QI (or its delegate) discretion,
* Current substance use disorders (DSM-V) (excluding tobacco and caffeine),
* History of, or current neurological illnesses, that would prevent participation in the trial,
* Current use or use during the previous month of antipsychotic medications,
* Learning disability, amnesia or other conditions that impede memory and attention,
* Visual impairments that prevent participation in the study,
* Personal or family history of schizophrenia, or psychosis (or psychosis-related) disorders,
* Antibiotic use in the last 4 weeks,
* Previous bariatric surgery,
* Current use or use in the past month of other weight-loss pharmaceuticals,
* Cannabis use in last 6 months,
* Known sensitivity to cannabis or other cannabinoid agents,
* Pregnancy or lactation (females), and
* For the optional imaging component of the study:

  * Presence of metal implants or objects unsafe for MRI such as cardiac pacemakers, metal fragments in the eye, and aneurysm clips in your brain
  * Piercings or jewelry that are unable to be removed
  * Tattoos inked with metal dyes

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Number of SAEs per treatment arm | 12 weeks of treatment
  Number of SAEs collected to assess nabilone safety
Number of dropouts per treatment arm | 12 weeks of treatment
  Number of dropouts collected to assess feasibility of study design and intervention

SECONDARY OUTCOMES:
Body weight | Baseline, then weekly for 12 weeks of treatment
  Change in body weight
Abdominal fat | One scan at baseline and one scan at Week 12
  Change in abdominal fat, as measured by abdominal MRI
Blood glucose levels | Blood drawn at baseline, Week 5, Week 9, and Week 12
  Change in metabolic biomarker (blood levels of glucose)
Blood insulin levels | Blood drawn at baseline, Week 5, Week 9, and Week 12
  Change in metabolic biomarker (blood levels of insulin)
Blood triglyceride levels | Blood drawn at baseline, Week 5, Week 9, and Week 12
  Change in metabolic biomarker (blood triglyceride levels)
Blood cholesterol levels | Blood drawn at baseline, Week 5, Week 9, and Week 12
  Change in metabolic biomarker (blood levels of HDL and LDL)
Blood leptin levels | Blood drawn at baseline, Week 5, Week 9, and Week 12
  Change in hunger-related hormones (blood levels of leptin)
Blood ghrelin levels | Blood drawn at baseline, Week 5, Week 9, and Week 12
  Change in hunger-related hormones (blood levels of ghrelin)
Blood PYY levels | Blood drawn at baseline, Week 5, Week 9, and Week 12
  Change in hunger-related hormones (blood levels of PYY)
Gut microbiota | Baseline, Week 12
  Stool samples collected for quantification of gut microbiome composition
Neural reactivity to food vs. control stimuli | Baseline, Week 12
  Task-based fMRI to determine differences in neural reactivity to food vs. control pictures

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada